CLINICAL TRIAL: NCT01517503
Title: Acceptance and Commitment Therapy vs. Cognitive Therapy for the Treatment of Major Depressive Disorder
Brief Title: Acceptance and Commitment Therapy Versus Cognitive Therapy for the Treatment of Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Paul M.G.Emmelkamp, Professor, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: METC 10/103
Record Dates: First submitted 2011-11-08; First posted 2012-01-25 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Cognitive Behavioral Therapy; Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Therapy (CT) (Experimental): Cognitive Therapy (CT)
  Interventions: Behavioral: Cognitive Therapy
- Acceptance and Commitment Therapy (ACT) (Experimental): Acceptance and Commitment Therapy (ACT)
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Cognitive Therapy — This interventions will target: (a) behavioral dysfunction, (b) situation-specific negative thinking and cognitive distortions, and (c) underlying dysfunctional beliefs or cognitions assumed to be related to the patient's current depression and risk of future depression. A maximum of 20 45-55 minute sessions will be provided, with sessions generally held weekly for the first 8 sessions and once every two weeks for the next 8 sessions.
  Other Names: Cognitive behavior therapy; cognitive behaviour therapy.
  Arms: Cognitive Therapy (CT)
Behavioral: Acceptance and Commitment Therapy — This interventions will use (a) acceptance, (b) commitment, (c) mindfulness, and (d) behavior change processes to produce reduction of depressive symptoms. A maximum of 20 45-55 minute sessions will be provided, with sessions generally held weekly for the first 8 sessions and once every two weeks for the next 8 sessions.
  Other Names: Mindfulness-based interventions
  Arms: Acceptance and Commitment Therapy (ACT)

SUMMARY:
The study will investigate the effectiveness of Cognitive Therapy and Acceptance and Commitment Therapy in a randomized controlled trial among patients with Major Depressive Disorder in routine clinical practice. Furthermore, the study will investigate whether each specific treatment approach is mediated by its proposed theoretical mechanism.

DETAILED DESCRIPTION:
The current study aims at investigating the effectiveness of Cognitive Therapy and Acceptance and Commitment Therapy in a randomized controlled trial among patients with MDD in routine clinical practice. Further, the study will investigate whether each specific treatment approach is mediated by its proposed theoretical mechanism. Patients have to meet diagnostic criteria for nonpsychotic MDD as determined by the Structured Interview for DSM-IV. Each client will receive either Cognitive Therapy or Acceptance and Commitment Therapy that will last between 16 to 20 sessions. Based on previous results, it is expected that both treatment forms will prove beneficial for the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting DSM-IV criteria for MDD
2. Between the ages of 18 and 65-years-old
3. Having sufficient fluency in Dutch to complete treatment and research protocol

Exclusion Criteria:

1. DSM-IV criteria for bipolar disorder (past or present)
2. Psychotic disorders
3. Substance dependence disorders (current or within the past 6 months), or
4. Organic brain syndrome.
5. Borderline or antisocial personality disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
QUICK INVENTORY OF DEPRESSIVE SYMPTOMATOLOGY (QIDS-SR) | pre-treatment, post-treatment, 6 and 12 months follow-up
  Change from pre-treatment to post-treatment, 6 months follow-up and 12 months follow-up
Hamilton Rating Scale for Depression | pre-treatment, post-treatment
  Change from pre-treatment to post-treatment.

SECONDARY OUTCOMES:
Decentering subscale of the Experiences Questionnaire | Pre-treatment, in-treatment, and 6 and 12 months follow-up.
  Change between sessions and to follow-up.
Acceptance and Action Questionnaire | Pre-treatment, in-treatment, and 6 and 12 months follow-up.
  Change between sessions and to follow-up.
Dysfunctional Attitude Scale-revised | Pre-treatment, in-treatment, and 6 and 12 months follow-up
  Change between sessions to follow-up.
Working Alliance Inventory | 3. session
Eurohis Quality of Life Scale | Pre-, post-treatment, 6 and 12 months follow-up
  Change pre-treatment to post-treatment and to follow-up.
Relationship Scales | Pre-, post-treatment, 12 months follow-up
  Change pre-treatment to post-treatment and to follow-up.
Implicit Attitude Test | Pre- and posttreatment
  Change pre-treatment to post-treatment
Structured Clinical Interview for DSM-IV (Major Depression Module) | Pre-treatment and post-treatment.
  Change in diagnosis of Major Depression Disorder from pre-treatment to post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Paul MG Emmelkamp, PhD, Principal Investigator — University of Amsterdam; Nexhmedin Morina, PhD, Study Director — University of Amsterdam
Locations (1):
- PsyQ, Zaandam, Netherlands

REFERENCES:
- [Derived] A-Tjak JGL, Morina N, Topper M, Emmelkamp PMG. One year follow-up and mediation in cognitive behavioral therapy and acceptance and commitment therapy for adult depression. BMC Psychiatry. 2021 Jan 14;21(1):41. doi: 10.1186/s12888-020-03020-1. PMID 33446152
- [Derived] A-Tjak JGL, Morina N, Boendermaker WJ, Topper M, Emmelkamp PMG. Explicit and implicit attachment and the outcomes of acceptance and commitment therapy and cognitive behavioral therapy for depression. BMC Psychiatry. 2020 Apr 7;20(1):155. doi: 10.1186/s12888-020-02547-7. PMID 32264845